CLINICAL TRIAL: NCT06242431
Title: Comparison of Serratus Posterior Superior Intercostal Plane Block (SPSIPB) and Pectoralis Nerve Block (PECS-II) Applications in the Treatment of Acute Pain After Coronary Artery Bypass Surgery (CABG)
Brief Title: Effects of Serratus Posterior Superior Intercostal Plane Block and Pectoralis Nerve Block in Coronary Artery Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Güvenç Doğan, Associated Professor, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-182
Record Dates: First submitted 2024-01-08; First posted 2024-02-05 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Postoperative;Pain Management
Keywords: CABG; Sternotomy; Pectoralis nerve block; Serratus posterior superior intercostal plane block

STUDY DESIGN:
Intervention Model Description: SPSIPB; The procedure will be carried out with the patient in the lateral decubitus position. After gently shifting the scapula laterally, the US probe is held sagittally at the upper corner of the scapula, and the 3rd rib and serratus posterior superior muscle are visualized. The block needle will be advanced in the cranio-caudal direction to enter between the serratus posterior superior and the 3rd rib. After confirming the block site, 30 ml of 0.25% concentration of marcaine (bupivacaine) will be used.
  PECS II; The block will be performed in the supine position of the patient, just anterior to the axillary line at the level of the 4th rib. After visualizing the serratus anterior, pectoralis major, and pectoralis minor muscles along with the ribs and pleura, the needle will be directed in-plane from cranial to caudal into the fascia of the serratus anterior muscle. Subsequently, 30 ml of bupivacaine with a 0.25% concentration will be applied.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group pectoralis nerve block (PECS-II) (Active Comparator): PECS II; The block will be performed in the supine position of the patient, just anterior to the axillary line at the level of the 4th rib. After visualizing the serratus anterior, pectoralis major, and pectoralis minor muscles along with the ribs and pleura, the needle will be directed in-plane from cranial to caudal into the fascia of the serratus anterior muscle. Subsequently, 30 ml of bupivacaine with a 0.25% concentration will be applied.
  Interventions: Procedure: Group pectoralis nerve block (PECS-II)
- Group serratus posterior superior intercostal plane block (SPSIPB) (Active Comparator): SPSIPB; The procedure will be carried out with the patient in the lateral decubitus position. After gently shifting the scapula laterally, the US probe is held sagittally at the upper corner of the scapula, and the 3rd rib and serratus posterior superior muscle are visualized. The block needle will be advanced in the cranio-caudal direction to enter between the serratus posterior superior and the 3rd rib. After confirming the block site, 30 ml of 0.25% concentration of marcaine (bupivacaine) will be used.
  Interventions: Procedure: Group serratus posterior superior intercostal plane block (SPSIPB)

INTERVENTIONS:
Procedure: Group serratus posterior superior intercostal plane block (SPSIPB) — SPSIPB; The procedure will be carried out with the patient in the lateral decubitus position. After gently shifting the scapula laterally, the US probe is held sagittally at the upper corner of the scapula, and the 3rd rib and serratus posterior superior muscle are visualized. The block needle will be advanced in the cranio-caudal direction to enter between the serratus posterior superior and the 3rd rib. After confirming the block site, 30 ml of 0.25% concentration of marcaine (bupivacaine) will be used.
  Arms: Group serratus posterior superior intercostal plane block (SPSIPB)
Procedure: Group pectoralis nerve block (PECS-II) — PECS II; The block will be performed in the supine position of the patient, just anterior to the axillary line at the level of the 4th rib. After visualizing the serratus anterior, pectoralis major, and pectoralis minor muscles along with the ribs and pleura, the needle will be directed in-plane from cranial to caudal into the fascia of the serratus anterior muscle. Subsequently, 30 ml of bupivacaine with a 0.25% concentration will be applied.
  Arms: Group pectoralis nerve block (PECS-II)

SUMMARY:
Postoperative analgesia is a critical risk factor for the development of pulmonary and cardiovascular complications in all types of chest surgery, particularly coronary artery bypass graft (CABG) surgery. Patients with high levels of pain who cannot breathe effectively may experience atelectasis, cardiac ischemia, and arrhythmias. This prolongs hospitalization and increases the frequency of postoperative pulmonary complications and morbidity. If postoperative acute pain is not adequately treated, it may lead to the development of chronic pain, hindering patients from recovering normal activities for an extended period. In addition to medications, various neuroaxial and peripheral nerve blocks can be used in cardiac surgery.

The use of high-dose heparin during surgery, along with neuroaxial anesthesia (thoracic epidural and intrathecal opioids), is controversial. Thoracic paravertebral block (TPVB) has demonstrated efficacy and is considered a method with fewer potential side effects compared to thoracic epidural anesthesia. However, TPVB has become less preferred in cardiac surgery due to its sympathetic blockade. Recently, peripheral nerve blocks have gained popularity as alternatives. These blocks include pectoralis nerve blocks (PECS-I, PECS-II), serratus anterior plane block (SAPB), serratus posterior superior intercostal plane block (SPSIPB), erector spinae plane block (ESPB), transverse thoracic plane blocks (TTMP), pectointercostal-fascial blocks (PIF), and intercostal nerve blocks. These blocks are newer and more superficially located compared to TPVB. Additionally, these fascial blocks are considered safer in terms of side effects as they do not cause sympathetic blockade like TPVB.

The hypothesis of this study is that SPSIPB can provide more extensive dermatomal analgesia compared to PECS-II, resulting in more effective postoperative analgesia. Therefore, this study plans to compare the analgesic effects of ultrasound-guided SPSIPB and PECS-II block applications in patients undergoing coronary artery bypass surgery with sternotomy.

DETAILED DESCRIPTION:
In many open cardiovascular operations, median sternotomy remains the most commonly used incision method due to its excellent visibility. This incision, made at the midline of the sternum, is frequently employed in open cardiovascular surgeries, resection of anterior mediastinal masses, radical thymectomies, and dissection of the superior mediastinum. The patient is placed in a supine position, and an incision is made at the midline of the sternum, starting from the jugular notch and extending to 1-2 cm below the xiphoid, ending on the linea alba. After passing through the subcutaneous tissue with an electrocautery, the anterior sternal fascia is reached, as there is no muscle tissue in the midline immediately after subcutaneous passage. Upon passing through the subcutaneous tissue with an electrocautery in the jugulum region, the clavicular heads of the clavioclavicular ligament, connecting the manubrium's undersurface, can be palpated. This ligament is cut and opened using electrocautery. The posterior surface of the sternum is dissected and separated from mediastinal structures by blunt dissections, starting from the posterior jugulum and below the xiphoid, using fingers. Subsequently, the midline of the sternum is marked with an electrocautery. An automatic saw is placed from the jugulum to the posterior surface of the sternum, and it is cut upwards slightly to avoid injuring the structures behind the sternum along the midline. After gentle retraction, the edges of the periosteum are cauterized at periosteal bleeding points, and hemostasis is achieved by applying bone wax. The sternal retractor is placed on the lower 2/3 of the sternum, minimizing the risk of occult fractures, neurological deficit, and damage to the innominate vein due to excessive tension on the superior costae. As the sternal retractor is slowly opened, access to the mediastinum is gained. Before closing the sternum at the end of the surgery, one or two chest tubes should be placed in the mediastinum or pleural spaces, depending on the need, for drainage. When closing the sternum, 4-7 thick stainless steel wires (no:5-6) are used, individually or in a crossed manner, to be securely fastened by tightly bending the wire ends at the midline, and the joined end is buried in the sternal tissue. Pectoral fascia and subcutaneous tissue are closed with absorbable sutures. Tight closure of the fascia on the sternum is crucial to prevent external contamination, infection, or clot collection. Postoperative pain after cardiac surgery is highly focused. Sternotomy, sternal retraction, internal mammary artery dissection, posterior rib dislocation or fracture, possible brachial plexus injury, mediastinal and pleural drains, saphenous vein damage all contribute to postoperative pain. In some patients, if the lateral decubitus position is required, position-related pain may develop in the shoulder joint. There is also a change in pain modulation in the peripheral and central nervous systems during the postoperative period. Opioid-based analgesia is associated with negative effects such as nausea, vomiting, sedation, urinary retention, itching, respiratory depression, and delayed extubation. Another analgesia method is the application of a thoracic epidural catheter. Thoracic epidural analgesia (TEA) can provide excellent "opioid-free" analgesia after cardiac surgery and is associated with a reduction in respiratory complications, arrhythmias, and mortality. However, in TEA, there is an increased risk of developing epidural hematoma during the perioperative period compared to non-cardiac surgeries due to the use of anticoagulant and antiplatelet agents in planned cardiac surgeries. Analgesia provided by serratus anterior plane block and pectoral muscle plane block does not cover the midline sternotomy pain. However, ultrasound-guided serratus posterior superior block (SPSPB), is a new interfascial plane block that has started to be routinely used for analgesia after invasive operations such as sternotomy. It relies on the injection above the serratus posterior superior muscle at the level of the 2nd or 3rd rib. This block provides analgesia in conditions such as interscapular pain, chronic myofascial pain syndromes, scapulocostal syndrome, and shoulder pain. The serratus posterior superior (SPS) muscle is located at the C7-T2 level and attaches to the lateral edges of the second and fifth ribs. It is innervated by the lower cervical and upper intercostal nerves. Analgesia is achieved by blocking these nerves with SPS block. In a cadaver study observed that the spread of SPSPB was staining only in the 7-10th intercostal levels on the surface fascia of the trapezius muscle on the left side, without staining on the right side. There was also significant staining deep in the trapezius muscle on both sides. Romboid major was distinctly stained both superficially and deeply, while romboid minor was only deep-stained. Therefore, SPSPB will provide successful analgesia in procedures involving the thoracic region, such as chronic myofascial pain, breast surgery, chest surgery, sternotomy. Another highly effective regional anesthesia method with high postoperative analgesic efficacy after breast and sternotomy surgeries is pectoral blocks. Pectoral block (PECS block) was described as an alternative to paravertebral and epidural blocks for pain control after surgery in patients undergoing breast surgery. PECS block has two types: Type I is performed between the pectoralis major and minor with local anesthetic and can be applied in the placement of subpectoral prosthesis with breast expander. PECS Block Type II is an injection of local anesthetic between pectoralis minor and serratus anterior muscles in addition to PECS Block Type I. PECS Type II block is one of the regional anesthesia techniques routinely used for postoperative analgesia in sternotomy, mastectomy, and axillary lymph node excision. Despite being a regional and superficial block, PECS block is highly reliable and easy to apply in terms of side effects. Both SPSPB and PECS II block are peripheral block applications that are quite popular, effective, and routinely used in clinical practice for postoperative analgesia in surgeries such as sternotomy and mastectomy in the field of anesthesiology.

There is currently no study in the literature comparing SPSPB and PECS type 2 block for post-thoracotomy analgesia. The hypothesis of this study is that SPSIPB can provide more extensive dermatomal analgesia compared to PECS-II, resulting in more effective postoperative analgesia. Therefore, this study plans to compare and evaluate the analgesic effects of ultrasound-guided SPSIPB and PECS-II block applications in patients undergoing coronary artery bypass surgery with sternotomy.

ELIGIBILITY:
Inclusion Criteria:

* Will undergo CABG surgery
* The American Society of Anesthesiologists (ASA) physical classification is 1-2-3.
* The volunteer has read and accepted the consent form
* Body mass index (BMI) <35

Exclusion Criteria:

* The patient does not want to participate in the study
* Patients with BMI >35
* Patients with ASA 4-5
* Those who are allergic to the local anesthetic used and the specified analgesic drug
* Those who declare that they are during pregnancy and breastfeeding
* Having uncontrollable anxiety
* Those with neuromuscular disease and peripheral nerve diseaseThose who used high doses of opioid medication 3 days before surgery
* Widespread chronic pain, diabetes mellitus, hepatic and renal failure
* Infection at the peripheral block needle insertion site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Examination with Visual analog scale | 24 hours
  Determination of patients' post-operative pain level. The Visual analog scale (VAS), a method that converts the patient's pain perception into a numerical form, will be used to assess postoperative pain. VAS has a numerical scale ranging from 0 to 100 mm. The patient will rate the intensity of pain on a scale from 0, indicating no pain, to 100, representing the worst imaginable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit university, Çorum, Çorum, Turkey (Türkiye)